CLINICAL TRIAL: NCT06213558
Title: The Effect of Rectangular Versus Square Archwire on Maxillary Canine Retraction: A Split Mouth Randomized Controlled Trial
Brief Title: The Effect of Rectangular Versus Square Archwire on Maxillary Canine Retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Talaat, Ahmed Talaat Helmy Khalifa, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahmed-Talaat
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Canine Retraction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation of rectangular archwire on maxillary canine retraction (Active Comparator): Evaluation of rectangular archwire on maxillary canine retraction
  Interventions: Device: Rectangular and square striaght archwire technique
- Evaluation of square archwire on maxillary canine retraction (Active Comparator): Evaluation of square archwire on maxillary canine retraction
  Interventions: Device: Rectangular and square striaght archwire technique

INTERVENTIONS:
Device: Rectangular and square striaght archwire technique — The Effect of Rectangular Versus Square Archwire on Maxillary Canine Retraction

SUMMARY:
The Effect of Rectangular Versus Square Archwire on Maxillary Canine Retraction

DETAILED DESCRIPTION:
his split-mouth randomized clinical trial will be carried out to evaluate the effect of rectangular versus square archwire on maxillary canine retraction.

ELIGIBILITY:
Inclusion Criteria:

- Individuals in permanent dentition phase with Class II canine and molar relationship that requires extraction of maxillary first premolars.

Individuals that require absolute anchorage using mini-implant.

No previous orthodontic treatment.

Good oral health

Age: 16-22 years

Exclusion Criteria:

- Patients with skeletal asymmetries.

Patients with syndromes or dental anomalies.

Patients with previous orthodontic treatment.

Evidence of root resorption.

Any medication affecting orthodontic tooth movement.

Ages: 16 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of canine retraction | 3 months
  The digital models will be superimposed using 3rd ruguae area. For each model, the distal point of the canine will be marked and the distance between 2 points will be calculated. The amount of canine retraction per month will be calculated from the difference in the canine cusp position in the four models.
  The digital models will be superimposed using 3rd ruguae area. For each model, the distal point of the canine will be marked and the distance between 2 points will be calculated. The amount of canine retraction per month will be calculated from the difference in the canine cusp position in the four models.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ta Khalifa, Master, Principal Investigator — Mansoura University
Locations (1):
- Mansoura, Al Mansurah, Daqahlya, Egypt

IPD SHARING:
Plan to Share IPD: No